CLINICAL TRIAL: NCT04489537
Title: Phase 3 Study to Evaluate the Efficacy and Safety of Subcutaneous Marzeptacog Alfa (Activated) For On Demand Treatment and Control of Bleeding Episodes in Subjects With Hemophilia A or Hemophilia B, With Inhibitors: The Crimson 1 Study
Brief Title: Study of Coagulation Factor VIIa Marzeptacog Alfa (Activated) in Subjects With Hemophilia A or B
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision (not a safety decision)
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAA-304
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MarzAA (Experimental): Coagulation Factor VIIa variant, 60 µg/kg by subcutaneous route, administered on-demand during bleeding episodes for a maximum of 3 doses as needed for hemostasis
  Interventions: Biological: MarzAA
- Standard of Care (Active Comparator): Standard of care administered on-demand during bleeding episodes
  Interventions: Biological: MarzAA

INTERVENTIONS:
Biological: MarzAA — A cross over design to assess the efficacy of a dosing regimen of 60 µg/kg of MarzAA compared with standard of care for the treatment of bleeding episodes.

SUMMARY:
The purpose of the trial is to evaluate the safety and efficacy of MarzAA for on-demand treatment and control of bleeding episodes in hemophilia A or B patients with inhibitors compared with their standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital hemophilia A or B with inhibitors
* Male or Female, age 12 or older
* History of frequent bleeding episodes
* Affirmation of informed consent with signature confirmation and assent for children between ages 12 to 17 before any study related activities

Exclusion Criteria:

* Previous participation in a clinical trial evaluating a modified rFVIIa agent
* Received an investigational drug within 30 days or 5 half-lives or absence of clinical effect
* Known hypersensitivity to trial or related product
* Known positive antibody to FVII or FVIIa detected by central lab at screening
* Have a coagulation disorder other than hemophilia A or B
* Be immunosuppressed
* Significant contraindication to participate

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Bleeding episode treatment success | 24 hours after the first administration of study drug
  Proportion of bleeding events treated with MarzAA achieving hemostatic efficacy based on a four-point scale according to the Investigator's assessment compared with standard of care.

CONTACTS AND LOCATIONS:
Locations (43):
- United States (2):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
- Hematology Center after Prof. R. Yeolyan, Yerevan, Armenia
- JSC "K.Eristavi National Center of Experimental and Clinical Surgery", Tbilisi, Georgia
- Magyar Honvédség Egészségügyi Központ, Országos Haemophilia Központ, Budapest, Hungary
- India (8):
  - Nirmal Hospital, Gujrāt
  - K.L.E.S Dr. Prabhakar Kore Hospital and Medical Research Centre, Kārnād
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - K.J Somaiya Hospital and Research Centre, Mumbai
  - MCGM - Comprehensive Thalassemia Care, Pediatric Hematology-Oncology & BMT Centre, Mumbai
  - Sahyadri Specialty Hospital, Mumbai
  - Grant Medical Foundation, Ruby Hall Clinic, Pune
  - All India Institute of Medical Sciences, Rishikesh, Rishikesh
- Italy (4):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
- Malaysia (5):
  - Hospital Ampang, Ampang
  - Raja Perempuan Zainab II Hospital, Kota Bharu
  - Queen Elizabeth Hospital Malaysia, Kota Kinabalu
  - Hospital Tunku Azizah Kuala Lumpur, Kuala Lumpur
  - Tuanku Ja'afar Hospital, Seremban, Sungai Petani
- Mexico (3):
  - Instituto de Investigaciones Aplicada a la Neurociencia A.C., Durango
  - Instituto Nacional de Pediatria, Mexico City
  - Investigación e Innovación en Medicina Traslacional S.A.P.I. de C.V., Mexico City
- Korczowski Bartosz, Gabinet Lekarski, Rzeszów, Poland
- Russia (2):
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - Medis, Llc, Nizhny Novgorod
- Haemophilia Comprehensive Care Centre, Johannesburg, South Africa
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de Malaga, Málaga
- Taiwan (2):
  - Changhua Christian Hospital (CCH), Changhua
  - Taichung Veterans General Hospital, Taichung
- Turkey (Türkiye) (4):
  - Akdeniz University Medical Faculty Hospital, Antalya
  - Istanbul University Faculty of Medicine, Istanbul
  - Ege University Medical Faculty, Izmir
  - Özel Acibadem Adana Hastanesi, Seyhan
- Ukraine (3):
  - "Cherkasy Regional Oncological Dispensary of Cherkasy Regional Council", Regional Treatment and Diagnostic Center of Hematology, Cherkasy
  - "Kyiv City Clinical Hospital #9" of Executive Body of Kyiv City Council (Kyiv City State Administration), City Scientific-Practical Centre of Diagnostics and Treatment, Kyiv
  - "Institute of Blood Pathology and Transfusion Medicine of National Academy of Medical Sciences of Ukraine", Haematology Department, Lviv
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No